CLINICAL TRIAL: NCT04222621
Title: Xiamen Registry of Pregnant Women and Offspring (REPRESENT): A Population-based, Long-term Follow-up Database Linking Four Major Healthcare Data Platforms
Brief Title: Xiamen Registry of Pregnant Women and Offspring (REPRESENT)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Collaborators: Xiamen Health and Medical Big Data Center, Xiamen Health Commission (Unknown)
Responsible Party: Principal Investigator, Sun Xin, Professor and director of Chinese Evidence-based Medicine Center, West China Hospital
Other Study IDs: REPRESENT
Record Dates: First submitted 2019-12-27; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Pregnant Women; Registries
Keywords: Population-based healthcare database; Registry; Pregnant women and offspring; Longitudinal study
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women
  Interventions: Other: Pregnant women without intervention

INTERVENTIONS:
Other: Pregnant women without intervention — Pregnant women with those exposures of interest determined in specific research based on the registry

SUMMARY:
To improve the health of women and children under the background of Healthy China 2030, the investigators developed REPRESENT by establishing a pregnancy registry in Xiamen, a sub-provincial city of over four million residents in east China, based on the Maternal and Child Health Management Platform, and then linking to three other platforms, i.e. Residents Healthcare Management Platform, Primary Healthcare Management Platform, and Electronic Healthcare Records (EHR) Platform, which had been developed since 2006. The registry documented information and events about pregnant women from registration at their first trimester to postpartum, and includes the childhood follow up records. The registry not only enables longitudinal follow up of pregnant women and their offspring, but also expands the scope of database from pre-pregnancy exposures to long-term outcomes by data linkage.

During the past 11 years (January 2008 to March 2019), the REPRESENT has accumulated data concerning more than 700 thousands pregnancies. The data volume is substantial with over 800 variables being documented, and most variables are designed as structured fields. The disease categories and codes are standardized according to the International Classification of Diseases 10th Revision (ICD-10). The whole process of data access, data extraction, data processing and data analysis was conducted through an internal-only accessible server at Xiamen Health and Medical Big Data Center. All investigators cannot access sensitive information, are required to sign data confidentiality agreement and should obtain approval by the Xiamen Health and Medical Big Data Center and the Chinese Evidence-based Medicine Center.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who registered at the Maternal and Child Health Management Platform in Xiamen.

Exclusion Criteria:

* None.

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All pregnant women registered at the Maternal and Child Health Management Platform were enrolled.
Study Population: Pregnant women who registered at the Maternal and Child Health Management Platform in Xiamen.
Sampling Method: Probability Sample
Enrollment: 761194 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of pre-eclampsia | Up to 42 weeks
  Maternal systolic blood pressure ≥ 140 mmHg and (or) diastolic pressure ≥ 90 mmHg, accompanied by any one of the following: urinary protein ≥ 0.3g/24 h, or the ratio of urinary protein and creatinine ≥ 0.3, or random urine protein ≥ (+) if quantitative urine protein is not available; no proteinuria but with any damages of heart, lung, liver, kidney and other important organs, or with abnormal changes of blood system, digestive system and nervous system, or placenta fetus involvement, etc.
Incidence of eclampsia | Up to 42 weeks
  Tonic-clonic seizures (convulsions) in preeclampsia patients, including convulsions and coma, not due to pre-existing or organic brain disorders.
Incidence of gestational diabetes | Up to 32 weeks
  By oral glucose tolerance test between 24 and 28 gestational weeks (fasting glucose ≥5.1 mmol/L, 1-h glucose ≥10.0 mmol/L, 2-h glucose ≥8.5 mmol/L; one abnormal result sufficient).
Incidence of ruptured uterus | Up to 42 weeks
  Rupture of maternal uterus confirmed by laparotomy.
Incidence of postpartum hemorrhage | Within 24h after delivery
  Postpartum bleeding volume ≥500 mL.
Incidence of maternal death | Up to 52 weeks
  Maternal death
Incidence of birth defects | Up to 7 years
  Birth defects such as anencephaly, spina bifida, encephalocele, hydrocephalus, cleft palate, cleft lip, microtia, esophageal atresia or stenosis, anorectal, hypospadias, ectropion of bladder, talipes equinovarus, polydactylism, ankylodactylia, congenital diaphragmatic hernia, umbilical cord prolapse, gastroschisis, conjoined twins, down syndrome, congenital heart disease, or other birth defects.
Incidence of preterm birth | Up to 37 weeks
  Delivery before 37th gestational weeks.
Incidence of neonatal birth weight | Up to 42 weeks
  Neonatal birth weight measured after birth.
Incidence of neonatal death | Within 28 days after delivery
  Neonatal death
Incidence of stillbirth | Up to 42 weeks
  Fetus death at or after 20-28 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, PhD, Study Director — Chinese Evidence-based Medicine Center, West China Hospital of Sichuan University

IPD SHARING:
Plan to Share IPD: Yes
Following the policy of Xiamen Health Commission, research institutions could apply for data access by submitting a formal study protocol, subjected to approval by the Xiamen Health and Medical Big Data Center and the Chinese Evidence-based Medicine Center. Ethical review and research registration are mandatory for all studies.